CLINICAL TRIAL: NCT04661527
Title: Sarilumab Treatment In cytoKinE Storm Caused by Infection With COVID-19
Acronym: STRIKESARS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Sanofi (Industry); Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRIKESARS-COV; 2020-001255-40 (EudraCT Number)
Record Dates: First submitted 2020-09-10; First posted 2020-12-10 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 Drug Treatment
MeSH Terms: interventions — sarilumab

STUDY DESIGN:
Intervention Model Description: Phase II, one-arm, open label, multicentric study, to evaluate treatment of severe COVID-19 with sarilumab prior to entry into the intensive care unit (ICU)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sarilumab arm (Experimental)
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Treatment with Sarilumab 200 mg IV x 2 doses 24 hours apart for first 5 patients. If no severe AE and no significant improvement within 48 hours, the dose will be increased for subsequent patients to 400 mg IV for the first dose and 200 mg or 400 mg IV for the second dose 24 hours later. Te second dose will be decided at the investigators discretion.
  Other Names: Kevzara®

SUMMARY:
Phase II, one-arm, open label, multicentric study, to evaluate treatment of severe COVID-19 with sarilumab prior to entry into the intensive care unit (ICU).

DETAILED DESCRIPTION:
Phase II, one-arm, open label, multicentric study, to evaluate treatment of severe COVID-19 with sarilumab prior to entry into the intensive care unit (ICU).

The primary objective of the trial is to evaluate the impact of sarilumab on the progression of COVID 19-associated respiratory failure as measured by the change in a severity rating on a 7-point severity index. Secondary objectives include the evaluation of safety of the drug and the assessment of the impact of Sarilumab on markers of systemic inflammation and the coagulation cascade, on mortality, and on oxygenation.

The trial has two phases. Firstly, patients with pneumonia in the setting of COVID-19 who meet inclusion criteria and have no exclusion criteria will be treated with 2 doses of 200 mg IV of Sarilumab in 24 hours. After internal review, if no AE are detected and if there is no significant improvement, the next 55 patients will be treated with two doses of 400 mg IV in 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performing study procedures. Oral consent will be accepted in order to avoid paper handling. Written consent by patient or representatives will be obtained as soon as possible.

   In the case of a vital emergency without the possibility of prior consent, a patient may be included in the study if the recommendations of the legislation are followed (RD 1090/2015, article 7), as stated in section 10.3 of the protocol.
2. Patient must be, in the investigator opinion, able to comply with all the protocol procedures.
3. Negative pregnancy test in case of fertile women*
4. Age >= 18
5. Infection by COVID-19 confirmed by rtPCR or other validated tests
6. Hospitalized (or documentation of a plan to admit to the hospital if the patient is in the emergency department) with illness of any duration, with evidence of pneumonia, and severe disease as defined by at least one of the following:

   1. High oxygen requirements (face mask with reservoir, non-invasive mechanical ventilation or high flow nasal cannula)
   2. Lymphocytes < 0.8 x 109/L
   3. Serum ferritin > 300ng/mL
   4. Increased levels of D-dimer (> 1500 ng/mL) or D-dimer progressively increasing (over 3 consecutive measurements) and reaching ≥ 1000 ng/mL.
   5. CPR > 10 mg/dL, or increasing over 24 hours

Exclusion Criteria:

Patients with any of the following exclusion criteria could not be included in the trial:

1. Hypersensitivity to the active substance or any of the excipients listed in section 6
2. Treatment with anti-IL 6, anti-IL-6R antagonists, or with Janus kinase inhibitors (JAKi) in the past 30 days
3. Alkylating agents including cyclophosphamide (CYC) within 6 months of baseline
4. Cyclosporine (CsA), azathioprine (AZA) or mycophenolate mofetil (MMF) or leflunomide within 4 weeks of baseline.
5. Alkylating agents including cyclophosphamide (CYC) within 6 months of baseline
6. Tumor necrosis factor (TNF) inhibitors within 2-8 weeks (etanercept within 2 weeks, infliximab, certolizumab, golimumab, or adalimumab within 8 weeks), or after at least 5 half-lives have elapsed, whichever is longer.
7. Intravenous immunoglobulin (IVIG) within the past 5 months or plans to receive during the study period
8. Current use of chronic oral corticosteroids for a non-COVID-19-related condition in a dose higher than prednisone 10 mg or equivalent per day
9. Current treatment with conventional synthetic disease-modifying antirheumatic drugs (DMARDs)/immunosuppressive agents
10. Patients who have received immunosuppressive antibody therapy within the past 5 months, including intravenous immunoglobulin
11. AST/ALT values > 5 x normal.
12. Neutropenia (< 0.5 x 109/L).
13. Sever thrombocytopenia (< 50 x 109/L).
14. Sepsis caused by an alternative pathogen.
15. Diverticulitis with risk of perforation.
16. Ongoing infectious dermatitis.
17. Patients with another active infection, including localized infections.
18. Pregnant or breast-feeding females will be excluded
19. Positive serology for following infection: HIV, Hepatitis B, or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in a severity rating on a 7-point ordinal scale | 15 days
  Impact of sarilumab on the progression of COVID-19 associated respiratory failure. A significant improvement in a 7-point severity index is anticipated to occur with treatment with sarilumab.

SECONDARY OUTCOMES:
Percentage of patients reporting each severity rating on a 7-point severity ordinal scale | 28 days
  Proportion of patients in each severity category at the end fo follow-up
Duration of mechanical ventilation | 28 days
  Duration of mechanical ventilation measured by days of ventilation since treatment
Evaluate the safety of sarilumab in patients with severe pneumonia caused by COVID 19 | 28 days
  All adverse events will be recorded in the CRF.
  Adverse Event is defined as any event that results in worsening of the health of the subject of the clinical trial, regardless of relationship to the experimental therapy. It can be any symptom, sign, illness or experience, including abnormal results of diagnostic procedures, that develops or worsens in severity during the course of the study.
  Serious Adverse Event are defined as any AE that is:
  * Fatal
  * Life-threatening*
  * Requires or prolongs hospital stay
  * Results in persistent or significant disability or incapacity
Number of ventilator free days in the first 28 days | 28 days
  Number of ventilator free days in the first 28 days
Patients requiring mechanical ventilation | 28 days
  Number and proportion of patients requiring mechanical ventilation
Change from baseline in PaO2/FiO2 in patients on mechanical ventilation | since day of intubation until day of extubation or up to day 28
  PaO2/FiO2 will be measured daily until extubation or day 28.
Time to improvement in oxygenation for at least 48 hours | 28 days
  Increase in SpO2/FiO2 of 50 or more compared to nadir SpO2/FiO2
Time to saturation > 93.9% on room air | 28 days
  Improvement on oxygenation using a threshold of SaO2 of 94% or better when breathing room air as a sign of improvement.
Time to resolution of fever without antipyretics for at least 48 hours (Tº > 36.6ºC - axilla; > 37.2ºC -oral; > 37.8 -rectal or tympanic) | 28 days
  Resolution of fever.
Changes from baseline in white blood cell count if available on V2, V3, V4, V5, and V6 | 28 days
  Changes in white blood count on visits number 2, 3 ,4, 5 and 6.
Changes from baseline in hemoglobin levels if available on V2, V3, V4, V5, and V6 | 28 days
  Changes in hemoglobin on visits number 2, 3 ,4, 5 and 6.
Changes from baseline in platelet cell count if available on V2, V3, V4, V5, and V | 28 days
  Changes in platelet counts on visits number 2, 3 ,4, 5 and 6.
Changes from baseline in D-Dimer leves if available on V2, V3, V4, V5, and V6 | 28 days
  Changes in D-dimer levels on visits number 2, 3 ,4, 5 and 6.
Number of deaths due to any cause | 28 days
  All-cause mortality
Organ failure | 28 days
  Events of organ failure after treatment: DIC, cardiac, hepatic, renal, cardiovascular
Changes from baseline in C Reactive protein if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates improvement or worsening of inflammation.
Changes from baseline in Ferritin leves if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates improvement or worsening of inflammation.
Changes from baseline in Troponin leves if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates potential myocardial involvement.
Changes from baseline in blood urea nitrogen leves if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates improvement or worsening of renal function
Changes from baseline in creatinine leves if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates improvement or worsening of renal function
Changes from baseline in blilirrubin leves if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates improvement or worsening of liver function
Changes from baseline in Aspartate transaminase (AST) leves if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates improvement or worsening of liver function
Changes from baseline in Alanine transaminase (ALT) leves if available on V2, V3, V4, V5, and V6 | 28 days
  Indicates improvement or worsening of liver function

CONTACTS AND LOCATIONS:
Overall Officials: Javier J Zulueta, MD, Principal Investigator — Clinica Universidad de Navarra
Locations (2):
- Spain (2):
  - Clínica Universidad de Navarra, Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Infanta Leonor, Madrid

IPD SHARING:
Plan to Share IPD: Undecided